CLINICAL TRIAL: NCT04898361
Title: Electrophysiological and Echocardiographic PREDICTors of Atrial Fibrillation Following Interventional Closure of Patent Foramen Ovale in Cryptogenic Stroke: PREDICT-AF-PFO
Brief Title: PFO Occlusion and Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Saarland (Other)
Responsible Party: Principal Investigator, Christian Ukena, Head of cardiac electrophysiology department, University Hospital, Saarland
Organization: Universität des Saarlandes (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREDICT-AF PFO
Record Dates: First submitted 2020-09-13; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Atrial Fibrillation New Onset; Embolic Stroke of Undetermined Source; Patent Foramen Ovale
MeSH Terms: conditions — Foramen Ovale, Patent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PFO closure (Active Comparator): Patients with embolic stroke of undetermined source (ESUS) with patent foramen ovale (PFO) eligible for interventional PFO occlusion receiving a structured electrophysiological study due to palpitations before the PFO closure. Extensive cardiac monitoring.
  Interventions: Procedure: PFO closure
- NO PFO (No Intervention): Patients with embolic stroke of undetermined source (ESUS) with NO patent foramen ovale (PFO) receiving a structured electrophysiological study due to palpitations. Extensive cardiac monitoring.

INTERVENTIONS:
Procedure: PFO closure — Interventional closure of a patent foramen oval preceded by an electrophysiological study
  Arms: PFO closure

SUMMARY:
Interventional closure of patent foramen ovale (PFO) associates with reduced risk of stroke recurrence in patients with cryptogenic ischemic stroke as reported in the recent CLOSE and REDUCE trials. The long-term follow-up results of the RESPECT and DEFENSE-PFO trial confirmed these findings. PFO closure is therefore recommended in patient with cryptogenic ischemic stroke and PFO according to the current German interdisciplinary guidelines. It is likely that the number of PFO closure procedures will increase significantly in the near future. However, new onset atrial fibrillation (AF) appears to increase in patients following this procedure. In the REDUCE study, new onset atrial fibrillation was detected in 6.6% patients in the PFO closure group compared with 0.4% in the control group (medical treatment); 59% of these patients were diagnosed within the first two weeks following the procedure and 83% within 45 days, respectively. These results were consistent with the CLOSE study: AF was detected in 4.6% patients in the intervention group vs. 0.9% in the control group. Up until today, markers to identify and quantify the individual risk of AF onset are lacking. Furthermore, under-reporting and under-detection of AF occurrence after PFO closure is likely. This study is designed to to assess the prevalence and and identification of electrophysiological and echocardiographic parameters of new-onset AF.

ELIGIBILITY:
Inclusion Criteria:

* Previous embolic stroke with undetermined source with…
* palpitations with clinical indication for an electrophysiological study (control group)
* PFO and clinical indication for interventional PFO closure according to current guidelines (intervention group)
* Sinus rhythm at time of inclusion with no history of AF
* Planned EP study due to reported palpitations or documented burden of non-sustained atrial arrythymias (>100 atrial ectopic beats /24 hours, atrial tachycardia)
* Written informed consent

Exclusion Criteria:

* previously documented AF
* indication for therapeutic anticoagulation
* uncontrolled diabetes mellitus
* acute coronary syndrom or acute cardiac decompensation within the last 6 months before enrollment
* enrolled in another study
* BMI > 40 kg/m²
* patients who are pregnant of breastfeeding life expectancy < 6 months
* relevant peripheral artery disease
* substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change in baseline heart rhythm, e.g. new-onset atrial fibrillation | 1, 3, 6, 12 months
  Rate of detection of new-onset atrial fibrillation with Holter and loop recorder monitoring after electrophysiological study

SECONDARY OUTCOMES:
Relevance of atrial refractory periods and inducibility of atrial arrhythmias during the electrophysiological study | 1 month
  Atrial refractory periods are measured and atrial arrhythmias are induced during the electrophysiological study. Measurement: electrophysiological study, Unit of measure: Rate of patients with induced AF during stimulation
Relevance of atrial refractory periods and inducibility of atrial arrhythmias during the electrophysiological study | 3 months
  Atrial refractory periods are measured and atrial arrhythmias are induced during the electrophysiological study. Measurement: electrophysiological study, Unit of measure: Rate of patients with induced AF during stimulation
Relevance of atrial refractory periods and inducibility of atrial arrhythmias during the electrophysiological study | 6 months
  Atrial refractory periods are measured and atrial arrhythmias are induced during the electrophysiological study. Measurement: electrophysiological study, Unit of measure: Rate of patients with induced AF during stimulation
Relevance of atrial refractory periods and inducibility of atrial arrhythmias during the electrophysiological study | 12 months
  Atrial refractory periods are measured and atrial arrhythmias are induced during the electrophysiological study. Measurement: electrophysiological study, Unit of measure: Rate of patients with induced AF during stimulation
Change in left atrial morphology (LA volume index) following PFO closure | 1 month
  Assessment of the change in left atrial morphology and function (LA volume index) during follow-up. Measurement: echocardiography, Unit of measure: Assessment of LA volume index, physiologocal parameter
Change in left atrial function (LA strain) following PFO closure | 1 month
  Assessment of the change in left atrial function (LA strain) during follow-up. Measurement: echocardiography, Unit of measure: Assessment of LA strain, physiologocal parameter
Change in new-onset AF following PFO closure | 1 month
  Assessment of new-onset AF during follow-up. Measurement: ECG, Holter ECG
Change in left atrial morphology (LA volume index) following PFO closure | 3 months
  Assessment of the change in left atrial function (LA strain) during follow-up. Measurement: echocardiography, Unit of measure: Assessment of LA strain, physiologocal parameter
Change in left atrial function (LA strain) following PFO closure | 3 months
  Assessment of the change in left atrial function (LA strain) during follow-up. Measurement: echocardiography, Unit of measure: Assessment of LA strain, physiologocal parameter
Change in new-onset AF following PFO closure | 3 months
  Assessment of new-onset AF during follow-up. Measurement: ECG, Holter ECG
Change in left atrial morphology (LA volume index) following PFO closure | 6 months
  Assessment of the change in left atrial function (LA strain) during follow-up. Measurement: echocardiography, Unit of measure: Assessment of LA strain, physiologocal parameter
Change in left atrial function (LA strain) following PFO closure | 6 months
  Assessment of the change in left atrial function (LA strain) during follow-up. Measurement: echocardiography, Unit of measure: Assessment of LA strain, physiologocal parameter
Change in new-onset AF following PFO closure | 6 months
  Assessment of new-onset AF during follow-up. Measurement: ECG, Holter ECG
Change in left atrial morphology (LA volume index) following PFO closure | 12 months
  Assessment of the change in left atrial function (LA strain) during follow-up. Measurement: echocardiography, Unit of measure: Assessment of LA strain, physiologocal parameter
Change in left atrial function (LA strain) following PFO closure | 12 months
  Assessment of the change in left atrial function (LA strain) during follow-up. Measurement: echocardiography, Unit of measure: Assessment of LA strain, physiologocal parameter
Change in new-onset AF following PFO closure | 12 months
  Assessment of new-onset AF during follow-up. Measurement: ECG, Holter ECG

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum des Saarlandes, Homburg, Saarland, Germany

IPD SHARING:
Plan to Share IPD: No